CLINICAL TRIAL: NCT07378124
Title: Efficacy and Safety Comparison of Lumenless Lead Versus Stylet-driven Lead in Intraoperative Application of Left Bundle Branch Pacing Guided by Continuous Pacing Monitoring With S-V Dissociation as the Primary Outcome: A Non-inferiority, Multicenter, Prospective Randomized Controlled Trial
Brief Title: LLL vs. SDL for LBBP: A Non-inferiority RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No.2 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PJ-NBEY-KY-2026-014-01
Record Dates: First submitted 2026-01-17; First posted 2026-01-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Bradycardia; Conduction Block, Atrioventricular
MeSH Terms: conditions — Bradycardia; Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDL group (Experimental): Subjects will receive implantation of a stylet-driven active fixation ventricular lead during the Left Bundle Branch Pacing (LBBP) procedure.
  Interventions: Procedure: SDL implantation
- LLL group (Active Comparator): Subjects will receive implantation of a lumenless active fixaion ventricular lead during the Left Bundle Branch Pacing (LBBP) procedure.
  Interventions: Procedure: LLL implantation

INTERVENTIONS:
Procedure: SDL implantation — Implantation of an SDL during LBBP procedures guided by continuous pacing monitoring, with the presence of S-V dissociation serving as the criterion for confirming optimal LBB lead positioning.
  Arms: SDL group
Procedure: LLL implantation — Implantation of an LLL during LBBP procedures guided by continuous pacing monitoring, with the presence of S-V dissociation serving as the criterion for confirming optimal LBB lead positioning.
  Arms: LLL group

SUMMARY:
Left Bundle Branch Pacing (LBBP) has emerged as one of the most commonly used physiological pacing modalities in clinical practice. However, the key determinants of procedural success lie in the accurate intraoperative identification of proper LBB lead positioning and the prevention of cardiac perforation. Our previous research has established a methodology for Lumenless Lead (LLL) implantation under the guidance of continuous pacing monitoring, and this methodology has been further adapted for Stylet-driven Lead (SDL) implantation. The present study is designed as a multicenter, randomized controlled trial, aiming to compare the differences in efficacy and safety between LLL and SDL during LBBP procedures guided by continuous pacing monitoring, with the presence of S-V dissociation serving as the criterion for confirming optimal LBB lead positioning.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic sick sinus syndrome (SSS);
* Complete or advanced atrioventricular block (AVB);
* Patients with heart failure complicated by left bundle branch block (LBBB) and biventricular dyssynchrony;
* Patients with atrial fibrillation (AF) complicated by refractory rapid ventricular rate who are scheduled for atrioventricular node ablation and permanent pacemaker implantation;
* Other patients who meet the indications for dual-chamber pacemaker implantation as specified in current guidelines

Exclusion Criteria:

* Patients who are ineligible for transvenous cardiac pacemaker implantation due to anatomical abnormalities, infections, or other factors;
* Patients with existing implantable cardiac electronic devices (ICEDs);
* Patients who opt for right-sided venous access for any reason;
* Patients with an expected survival of less than 1 year;
* Patients who have been enrolled in other clinical trials related to implantable cardiac electronic devices within 3 months prior to enrollment in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2026-01-24 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint | During the LBBP procedure
  The primary efficacy endpoint is defined as the success rate of intraoperative implantation of the left bundle branch lead with the documentation of S-V dissociation.
The primary safety endpoint | From start of the procedure to the end of follow-up at 6 months
  The primary safety endpoint is defined as a composite endpoint consisting of the following anticipated procedure-related serious adverse events (SAEs).

SECONDARY OUTCOMES:
Procedural success rate | During the procedure.
  The procedural success rate, defined as completion of LBB lead implantation in the interventricular septum, meets the criteria for left bundle branch area pacing as defined in current guidelines. Although S-V dissociation is not achieved, at least two visualized indicators are observed when the pacing output is set at ≤2 V/0.5 ms.
Abnormal parameters detected during follow-up | From the start of procedure to the end of follow-up at 6 months
  Clinically significant abnormalities in pacing lead parameters detected during pacemaker programming throughout the follow-up period.
Assessment of cardiac function during follow-up | From the start of procedure to the end of follow-up at 6 months
  Postoperative occurrence of pacemaker-related heart failure or progression of pre-existing cardiac insufficiency.
Assessment of quality of life. | From the start of procedure to the end of follow-up at 6 months
  Changes in subjects' quality of life (assessed by the multipurpose short-form [SF-12] Health Survey Score). The SF-12 scale assesses eight health domains. Its standardized scores range from 0 to 100, and a higher total score indicates better overall health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo No.2 Hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shen J, Jiang L, Wu H, Cai X, Zhuo S, Pan L. A Continuous Pacing and Recording Technique for Differentiating Left Bundle Branch Pacing From Left Ventricular Septal Pacing: Electrophysiologic Evidence From an Intrapatient-Controlled Study. Can J Cardiol. 2023 Jan;39(1):1-10. doi: 10.1016/j.cjca.2022.09.008. Epub 2022 Sep 14. PMID 36113707
- [Result] Shen J, Jiang L, Wu H, Zhang L, Li H, Pan L. Electrophysiological characteristics of lead position-dependent electrogram uninterrupted transition during left bundle branch pacing. Heart Rhythm. 2025 May;22(5):1279-1288. doi: 10.1016/j.hrthm.2024.10.062. Epub 2024 Nov 6. PMID 39515497
- [Result] Wu H, Jiang L, Chen W, Zhuo S, Shen J, Zhang L, Zhang Y, Peng X. Short- to Mid-Term Efficacy and Safety of Left Bundle Branch Pacing Guided by Continuous Uninterrupted Paced Intracardiac Electrogram Monitoring Targeting Transition to Selective Left Bundle Branch Capture. J Cardiovasc Electrophysiol. 2025 Nov;36(11):2839-2848. doi: 10.1111/jce.70054. Epub 2025 Aug 19. PMID 40831032
- [Result] Shen J, Jiang L, Wu H, Li H. Continuous Pacing and Recording Technique: A Real-Time Feedback Approach for Left Bundle Branch Pacing. CJC Open. 2025 Jul 22;7(10):1357-1365. doi: 10.1016/j.cjco.2025.07.008. eCollection 2025 Oct. PMID 41180340